

### Clinical Development

## EGF816 (Nazartinib)

### CEGF816X2101 / NCT02108964

A Phase I/II, multicenter, open-label study of EGFRmut–TKI EGF816 administered orally in adult patients with EGFRmut solid malignancies

## Statistical Analysis Plan (SAP) for close-out CSR

Document type: SAP Documentation

Document status: Final

Release date: 16-May-2023

Number of pages: 15

Property of Novartis

Confidential

May not be used, divulged, published or otherwise disclosed without the consent of Novartis

Template Version 4.0, Effective from 23-Apr-2021

# Document History – Changes compared to previous final version of SAP

| Date | Time<br>point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| 16-May-<br>2023 | Prior to<br>DBL | Creation of final version | N/A - First version | NA |

#### **Table of contents**

| | Table of contents | 3 |
|---|---------------------------------------|---|
| | Introduction | |
| 2 | Planned tables, figures, and listings | 3 |

#### 1 Introduction

This statistical analysis plan (SAP) describes all planned analyses for the close-out clinical study report (CSR) of study CEGF816X2101, a phase I/II, multicenter, open-label study of EGFRmut-TKI EGF816 administered orally in adult patients with EGFRmut solid malignancies.

The close-out CSR will present the results of cumulative study data which are collected up to the LPLV date. The outputs planned for the close-out CSR will be a subset of the primary analysis outputs that need to be updated after the data cut-off date for the primary analysis. The list of outputs are specified in Section 2.

The statistical methods for the analyses in the final CSR, including data analysis general information, analysis of baseline characteristics, treatments and analysis supporting primary, secondary and exploratory objectives, will remain unchanged from that documented in the SAP for the primary analysis.

At the time of the finalization of the SAP, the following versions of study documents referred to are in place:

- [CEGF816X2101 SAP CSR 1 amendment3](dated 14-Jun-2018)
- [CEGF816X2101 TFL CSR addendum 1 0] (date 18-Oct-2018)

## 2 Planned tables, figures, and listings

The table below provides the list of outputs that need to be generated, with additional guidelines added under 'Programming notes'.

| Output number in close-out CSR | Output title in close-out CSR | Output number in primary analysis CSR | Output title in primary analysis CSR | Programming<br>Notes |
|---|---|---|---|---|
| Table 2-1 | Overview of<br>adverse events -<br>Phase I (Safety set) | Table 12-4a | Overview of adverse<br>events - Phase I<br>(Safety set) | |
| Table 2-2 | Overview of<br>adverse events -<br>Phase II (Safety<br>set) | Table 12-4b | Overview of adverse<br>events - Phase II<br>(Safety set) | |
| Table 2-3 | Adverse events by preferred term - Phase I (Safety set) | Table 12-5a | Adverse events by preferred term - Phase I (Safety set) | |

| Table 2-4 | Adverse events by preferred term - Phase II (Safety set) | Table 12-5b | Adverse events by preferred term - Phase II (Safety set) | |
|---|---|---|---|---|
| Table 2-5 | Overall survival -<br>Phase I (Full<br>analysis set) | Table 14.2-2.12a | Overall survival -<br>Phase I (Full analysis<br>set) | Prepared as cell-<br>based table to be<br>used as in-text. |
| Table 2-6 | Overall survival -<br>Phase II (Full<br>analysis set) | Table 14.2-2.12b | Overall survival -<br>Phase II (Full<br>analysis set) | Prepared as cell-<br>based table to be<br>used as in-text. |
| Table 14.1-1.1a | Subject disposition - Phase I (Full analysis set) | Table 14.1-1.1a | Subject disposition -<br>Phase I (Full analysis<br>set) | |
| Table 14.1-1.1b | Subject disposition - Phase II (Full analysis set) | Table 14.1-1.1b | Subject disposition -<br>Phase II (Full<br>analysis set) | |
| Table 14.1-1.3a | Protocol deviations - Phase I (Full analysis set) | Table 14.1-1.3a | Protocol deviations -<br>Phase I (Full analysis<br>set) | |
| Table 14.1-1.3b | Protocol deviations - Phase II (Full analysis set) | Table 14.1-1.3b | Protocol deviations -<br>Phase II (Full<br>analysis set) | |
| Table 14.1-3.1a | Demographics and<br>baseline<br>characteristics -<br>Phase I (Full<br>analysis set) | Table 14.1-3.1a | Demographics and<br>baseline<br>characteristics -<br>Phase I (Full analysis<br>set) | |
| Table 14.1-3.1b | Demographics and<br>baseline<br>characteristics -<br>Phase II (Full<br>analysis set) | Table 14.1-3.1b | Demographics and<br>baseline<br>characteristics -<br>Phase II (Full<br>analysis set) | |
| Table 14.1-3.9a | Antineoplastic therapy since discontinuation of study drug by ATC class and preferred term - Medication - Phase I (Full analysis set) | Table 14.1-3.9a | Antineoplastic therapy since discontinuation of study drug by ATC class and preferred term - Medication - Phase I (Full analysis set) | |
| Table 14.1-3.9b | Antineoplastic therapy since discontinuation of study drug by ATC class and preferred term - Medication - Phase II (Full analysis set) | Table 14.1-3.9b | Antineoplastic therapy since discontinuation of study drug by ATC class and preferred term - Medication - Phase II (Full analysis set) | |
| Table 14.2-1.4b | Progression-free<br>survival per BIRC<br>- Phase II (Full<br>analysis set) | Table 14.2-1.4b | Progression-free<br>survival per BIRC -<br>Phase II (Full<br>analysis set) | |

| Table 14.2-1.5b | Time to response<br>(CR+PR) as per<br>BIRC - Phase II<br>(Full analysis set) | Table 14.2-1.5b | Time to response<br>(CR+PR) as per<br>BIRC - Phase II<br>(Full analysis set) |
|---|---|---|---|
| Table 14.2-1.6b | Duration of<br>response (CR+PR)<br>as per BIRC -<br>Phase II (Full<br>analysis set) | Table 14.2-1.6b | Duration of response<br>(CR+PR) as per<br>BIRC - Phase II<br>(Full analysis set) |
| Table 14.2-2.4a | Progression-free<br>survival per<br>investigator<br>assessment - Phase<br>I (Full analysis set) | Table 14.2-2.4a | Progression-free<br>survival per<br>investigator<br>assessment - Phase I<br>(Full analysis set) |
| Table 14.2-2.4b | Progression-free<br>survival per<br>investigator<br>assessment - Phase<br>II (Full analysis<br>set) | Table 14.2-2.4b | Progression-free<br>survival per<br>investigator<br>assessment - Phase II<br>(Full analysis set) |
| Table 14.2-2.5a | Time to response<br>(CR+PR) as per<br>investigator -<br>Phase I (Full<br>analysis set) | Table 14.2-2.5a | Time to response<br>(CR+PR) as per<br>investigator - Phase I<br>(Full analysis set) |
| Table 14.2-2.5b | Time to response<br>(CR+PR) as per<br>investigator -<br>Phase II (Full<br>analysis set) | Table 14.2-2.5b | Time to response<br>(CR+PR) as per<br>investigator - Phase<br>II (Full analysis set) |
| Table 14.2-2.6a | Duration of<br>response (CR+PR)<br>as per investigator<br>- Phase I (Full<br>analysis set) | Table 14.2-2.6a | Duration of response<br>(CR+PR) as per<br>investigator - Phase I<br>(Full analysis set) |
| Table 14.2-2.6b | Duration of<br>response (CR+PR)<br>as per investigator<br>- Phase II (Full<br>analysis set) | Table 14.2-2.6b | Duration of response<br>(CR+PR) as per<br>investigator - Phase<br>II (Full analysis set) |
| Table 14.2-2.12a | Overall survival -<br>Phase I (Full<br>analysis set) | Table 14.2-2.12a | Overall survival -<br>Phase I (Full analysis<br>set) |
| Table 14.2-2.12b | Overall survival -<br>Phase II (Full<br>analysis set) | Table 14.2-2.12b | Overall survival -<br>Phase II (Full<br>analysis set) |
| Table 14.3-1.1a | Duration of<br>exposure to<br>EGF816 - Phase I<br>(Safety set) | Table 14.3-1.1a | Duration of exposure<br>to EGF816 - Phase I<br>(Safety set) |
| Table 14.3-1.1b | Duration of exposure to | Table 14.3-1.1b | Duration of exposure<br>to EGF816 - Phase II<br>(Safety set) |

| | ECEO16 DI II | I | | 1 |
|---|---|---|---|---|
| | EGF816 - Phase II | | | |
| | (Safety set) | | D CECEO16 | |
| T 11 142 12 | Dose of EGF816 | T 11 142 12 | Dose of EGF816 | |
| Table 14.3-1.2a | received - Phase I | Table 14.3-1.2a | received - Phase I | |
| | (Safety set) | | (Safety set) | |
| T 11 142 121 | Dose of EGF816 | T 11 142 121 | Dose of EGF816 | |
| Table 14.3-1.2b | received - Phase II | Table 14.3-1.2b | received - Phase II | |
| | (Safety set) | | (Safety set) | |
| | Dose adjustments | | Dose adjustments and | |
| Table 14.3-1.3a | and discontinuation of EGF816 - Phase | Table 14.3-1.3a | discontinuation of | |
| | | | EGF816 - Phase I | |
| | I (Safety set) | | (Safety set) | |
| | Dose adjustments and discontinuation | | Dose adjustments and discontinuation of | |
| Table 14.3-1.3b | of EGF816 - Phase | Table 14.3-1.3b | EGF816 - Phase II | |
| | II (Safety set) | | (Safety set) | |
| | Hematology shift table based on CTC | | Hematology shift table based on CTC | |
| Table 14.3-3.1a | grades - Phase I | Table 14.3-3.1a | grades - Phase I | |
| | (Safety set) | | (Safety set) | |
| | Hematology shift | | Hematology shift | |
| | table based on CTC | | table based on CTC | |
| Table 14.3-3.1b | grades - Phase II | Table 14.3-3.1b | grades - Phase II | |
| | (Safety set) | | (Safety set) | |
| | Hematology shift | | Hematology shift | |
| | table based on | | table based on normal | |
| Table 14.3-3.2a | normal ranges - | Table 14.3-3.2a | ranges - Phase I | |
| | Phase I (Safety set) | | (Safety set) | |
| | Hematology shift | | , , | |
| | table based on | | Hematology shift | |
| Table 14.3-3.2b | normal ranges - | Table 14.3-3.2b | table based on normal | |
| | Phase II (Safety | | ranges - Phase II | |
| | set) | | (Safety set) | |
| | Biochemistry shift | | Biochemistry shift | |
| T 11 142 22 | table based on CTC | T. 1.1. 1.4.2.2.2 | table based on CTC | |
| Table 14.3-3.3a | grades - Phase I | Table 14.3-3.3a | grades - Phase I | |
| | (Safety set) | | (Safety set) | |
| | Biochemistry shift | | Biochemistry shift | |
| Table 14.3-3.3b | table based on CTC | Table 14.3-3.3b | table based on CTC | |
| 1 4.3-3.30 | grades - Phase II | 1 able 14.3-3.30 | grades - Phase II | |
| | (Safety set) | | (Safety set) | |
| | Biochemistry shift | | Biochemistry shift | |
| Table 14.3-3.4a | table based on | Table 14.3-3.4a | table based on normal | |
| 1 4010 17.3-3.44 | normal ranges - | 1 4010 17.3-3.44 | ranges - Phase I | |
| | Phase I (Safety set) | | (Safety set) | |
| | Biochemistry shift | | Biochemistry shift | |
| | table based on | | table based on normal | |
| Table 14.3-3.4b | normal ranges - | Table 14.3-3.4b | ranges - Phase II | |
| | Phase II (Safety | | (Safety set) | |
| | set) | | ` ' | |
| Table 14.3-3.5a | Categorical | Table 14.3-3.5a | Categorical analysis | |
| | analysis of hepatic | - =================================== | of hepatic laboratory | |

| | 1-1 | | values - Phase I |
|---|---|---|---|
| | laboratory values - | | |
| | Phase I (Safety set) | | (Safety set) |
| Table 14.3-3.5b | Categorical<br>analysis of hepatic<br>laboratory values -<br>Phase II (Safety<br>set) | Table 14.3-3.5b | Categorical analysis<br>of hepatic laboratory<br>values - Phase II<br>(Safety set) |
| Table 14.3-4.1a | Vital signs shift<br>table based on<br>normal ranges -<br>Phase I (Safety set) | Table 14.3-4.1a | Vital signs shift table<br>based on normal<br>ranges - Phase I<br>(Safety set) |
| Table 14.3-4.1b | Vital signs shift<br>table based on<br>normal ranges -<br>Phase II (Safety<br>set) | Table 14.3-4.1b | Vital signs shift table<br>based on normal<br>ranges - Phase II<br>(Safety set) |
| Table 14.3-4.2a | Notable vital sign<br>values - Phase I<br>(Safety set) | Table 14.3-4.2a | Notable vital sign<br>values - Phase I<br>(Safety set) |
| Table 14.3-4.2b | Notable vital sign<br>values - Phase II<br>(Safety set) | Table 14.3-4.2b | Notable vital sign<br>values - Phase II<br>(Safety set) |
| Table 14.3-5.1a | Change from<br>baseline ECG<br>parameters by<br>timepoint - Phase I<br>(Safety set) | Table 14.3-5.1a | Change from baseline<br>ECG parameters by<br>timepoint - Phase I<br>(Safety set) |
| Table 14.3-5.1b | Change from baseline ECG parameters by timepoint - Phase II (Safety set) | Table 14.3-5.1b | Change from baseline<br>ECG parameters by<br>timepoint - Phase II<br>(Safety set) |
| Table 14.3-5.2a | Notable ECG<br>values - Phase I<br>(Safety set*) | Table 14.3-5.2a | Notable ECG values - Phase I (Safety set*) |
| Table 14.3-5.2b | Notable ECG<br>values - Phase II<br>(Safety set*) | Table 14.3-5.2b | Notable ECG values - Phase II (Safety set*) |
| Figure 14.3-1.1a | eDISH plot: Total<br>bilirubin vs<br>ALT/AST - Phase<br>I (Safety set) | Figure 14.3-1.1a | eDISH plot: Total<br>bilirubin vs<br>ALT/AST - Phase I<br>(Safety set) |
| Figure 14.3-1.1b | eDISH plot: Total<br>bilirubin vs<br>ALT/AST - Phase<br>II (Safety set) | Figure 14.3-1.1b | eDISH plot: Total<br>bilirubin vs<br>ALT/AST - Phase II<br>(Safety set) |
| Figure 14.3-1.2a | Individual subject<br>plot of ULN-<br>normalized LFT<br>values for subjects<br>with ALT>3xULN<br>or AST>3xULN or<br>Total Bilirubin>2x | Figure 14.3-1.2a | Individual subject plot of ULN-normalized LFT values for subjects with ALT>3xULN or AST>3xULN or Total Bilirubin>2x |

| ULN post-baseline - Phase I (Safety set) Individual subject plot of ULN-normalized LFT values for subjects with ALT>3xULN or Total Bilitrubin>2x ULN post-baseline - Phase II (Safety set) Table 14.3.1- 2a Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.3a Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Tab | | | 1 | TTT | T |
|---|---|---|---|---|---|
| Individual subject plot of ULN-normalized LFT values for subjects with ALT=3xULN or Total Bilirubin>2x ULN post-baseline - Phase II (Safety set) | | | | | |
| Individual subject plot of ULN-normalized LFT values for subjects with ALT-3xULN or AST>3xULN or Total Bilirubin>2x ULN post-baseline -Phase II (Safety set) | | ` • | | Phase I (Safety set) | |
| Figure 14.3-1.2b Adverse events by with ALT-3xULN or Adverse events by with ALT-3xULN or Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Figure 14.3-1.2b Adverse events by with ALT-3xULN or Adverse events by with AL | | | | | |
| Figure 14.3-1.2b Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Figure 14.3-1-2b Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Figure 14.3-1-2b Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set | | | | Individual subject | |
| Figure 14.3-1.2b Adverse events by System organ class, preferred term and maximum grade - Phase I (Safety set) Figure 14.3-1.2b Adverse events by System organ class, preferred term and maximum grade - Phase II (Safety set) Figure 14.3-1.2b Adverse events by System organ class, preferred term and maximum grade - Phase II (Safety set) Figure 14.3-1.2b Adverse events by System organ class, preferred term and maximum grade - Phase II (Safety set) Figure 14.3-1.2b Adverse events by System organ class, preferred term and maximum grade - Phase II (Safety set) Figure 14.3-1.2b Adverse events by System organ class, preferred term and maximum gr | | | | | |
| Figure 14.3-1.2b with ALTP-3xULN or AST>3xULN or AST>3xULN or AST>3xULN or Total Bilirubin>2x ULN post-baseline - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Table | | | | | |
| Figure 14.3-1.2b or AST>3xULN or Total Bilirubin>2x ULN post-baseline - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Tabl | | | | | |
| Table 14.3.1- 1.2a Table 14.3.1- 1.2b Table 14.3.1- 1.3a Table 14.3.1- 1.3b Table 14.3.1- Table 14.3.1 | Figure 14 3-1 2b | | Figure 14 3-1 2b | | |
| Total Bilirubin>2x ULN post-baseline Phase II (Safety set) | 118010 1110 1120 | | 118010 1110 1120 | | |
| ULN post-baseline - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Table 1 | | | | - | |
| Table 14.3.1- Table | | | | | |
| Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.2a Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.3a Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4a Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) | | , , | | | |
| Table 14.3.1- 1.2a system organ class, preferred term and maximum grade - Phase I (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.3b Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4a Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Adverse events | | , | | ` · | |
| Table 14.3.1- Ta | | | | | |
| 1.2a preferred term and maximum grade - Phase I (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- Table 14. | Table 14.3.1- | | Table 14.3.1- | | |
| Table 14.3.1- Ta | | | _ | | |
| Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.3a Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) | 1.2 | - C | 1.2 | $\mathbf{c}$ | |
| system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.3a Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Table 14.3.1- Ta | | | | Phase I (Safety set) | |
| Table 14.3.1- 1.2b | | _ | | Adverse events by | |
| Table 14.3.1- Table 14.3.1 | T 11 14 2 1 | | T 11 14 2 1 | • | |
| Table 14.3.1- Table 14.3.1 | | | | | |
| Table 14.3.1- 1.3a Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Adverse events | 1.2b | | 1.2b | | |
| Table 14.3.1- Ta | | - | | | |
| Table 14.3.1- 1.3a adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4b Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.5a Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.5a Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.5a Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.5a Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.5a Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.5a Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) | | , | | ` • | |
| Table 14.3.1- 1.3a System organ class, preferred term and maximum grade - Phase I (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.3b Table 14.3.1- 1.3a Table 14.3.1- 1.3a Table 14.3.1- 1.3a Table 14.3.1- 1.3a Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Table 14.3.1- 1.4b Table 14.3.1- 1.4b Table 14.3.1- 1.4b Table 14.3.1- 1.4b Table 14.3.1- 1.5a Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Table 14.3.1- 1.5a Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) | | | | | |
| 1.3a preferred term and maximum grade - Phase I (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.3b Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4a Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Adverse events | T 11 1401 | _ | T 11 1401 | _ | |
| Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Adverse events Table 14.3.1- 1.4b Adverse events | | | _ | | |
| Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Table 14.3.1- 1.4b Phase I (Safety set) Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Table 14.3.1- 1.4b Phase I (Safety set) Table 14.3.1- 1.4b Table 14.3.1- 1.4b Phase I (Safety set) Table 14.3.1- 1.4b Phase I (Safety set) Table 14.3.1- 1.4b Adverse events Adverse events | 1.3a | | 1.3a | | |
| Table 14.3.1- 1.3b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4a Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Treatment-related adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a Table 14.3.1- 1.4b Table 14.3.1- 1.4a Tabl | | | | | |
| Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Table 14.3.1- Adverse events Table 14.3.1- Adverse events Adverse events | | | | Phase I (Safety set) | |
| Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Table 14.3.1- 1.4b Table 14.3.1- Adverse events by system organ class, preferred term and maximum grade events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Table 14.3.1- Adverse events Table 14.3.1- Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) | | | | Treatment-related | |
| Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.3b Table 14.3.1- 1.4a Table 14.3.1- 1.4a Table 14.3.1- 1.4b Table 14.3.1- Adverse events Table 14.3.1- Adverse events Table 14.3.1- Adverse events Table 14.3.1- Adverse events | | • | | adverse events by | |
| 1.3b preferred term and maximum grade - Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4a | Table 14.3.1- | | Table 14.3.1- | • | |
| Table 14.3.1- Table 14.3.1- Table 14.3.1- 1.4a Table 14.3.1- Table 14.3.1- Adverse events Adverse events Adverse events | 1.3b | | 1.3b | | |
| Table 14.3.1- Adverse events Table 14.3.1- Table 14.3.1- Adverse events Adverse events Adverse events Adverse events Phase II (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events Adverse events Adverse events Adverse events | | | | | |
| Serious adverse events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- Table 14.3.1- Table 14.3.1- Table 14.3.1- Table 14.3.1- Table 14.3.1- Table 14.3.1- Adverse events Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Table 14.3.1- Adverse events Table 14.3.1- Table 14.3.1- Adverse events Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events Adverse events | | ` • | | | |
| Table 14.3.1- 1.4a events by system organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Table 14.3.1- 1.4a events by system organ class, preferred term and maximum grade - Phase I (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Table 14.3.1- Adverse events Table 14.3.1- Adverse events Fable 14.3.1- Adverse events Adverse events Adverse events | | | | Comous adverse | |
| Table 14.3.1- 1.4a organ class, preferred term and maximum grade - Phase I (Safety set) Table 14.3.1- 1.4b Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events Table 14.3.1- Table 14.3.1- Adverse events Table 14.3.1- Table 14.3.1- Adverse events Table 14.3.1- Adverse events Table 14.3.1- Adverse events Adverse events | | | | | |
| 1.4a preferred term and maximum grade - Phase I (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- 1.4b Adverse events Table 14.3.1- Table 14.3.1- Adverse events Table 14.3.1- Adverse events Table 14.3.1- Adverse events Table 14.3.1- Adverse events Table 14.3.1- Adverse events | Toble 1/1 2 1 | | Toble 1/1 2 1 | | |
| maximum grade - Phase I (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Table 14.3.1- Adverse events Table 14.3.1- Table 14.3.1- Adverse events Table 14.3.1- Adverse events Table 14.3.1- Adverse events Adverse events Adverse events | | | | | |
| Phase I (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Table 14.3.1- Adverse events (Safety set) Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events Adverse events Adverse events | 1. <del>4</del> a | | 1.44 | | |
| Table 14.3.1- 1.4b Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Adverse events Adverse events Adverse events Adverse events | | | | | |
| Table 14.3.1- 1.4b events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events Serious adverse events by system organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events Adverse events Adverse events | | ` . | | (Saicly Sel) | |
| Table 14.3.1- 1.4b organ class, preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events Table 14.3.1- Adverse events Table 14.3.1- Adverse events Adverse events | | | | | |
| Table 14.3.1- 1.4b preferred term and maximum grade - Phase II (Safety set) Table 14.3.1- Adverse events Table 14.3.1- Adverse events Adverse events Table 14.3.1- Adverse events | | 2 2 | | | |
| maximum grade - Phase II (Safety set) Table 14.3.1- Table 14.3.1- Table 14.3.1- Table 14.3.1- Table 14.3.1- Iterm and maximum grade - Phase II (Safety set) Adverse events Adverse events | | | | | |
| Phase II (Safety set) Table 14.3.1- Adverse events Table 14.3.1- Adverse events | 1.4b | | 1.4b | | |
| set) Salety set) Adverse events Table 14 3 1- Adverse events | | <u> </u> | | U | |
| Table 14 3 1- Adverse events Table 14 3 1- Adverse events | | | | (Safety set) | |
| Table 14 3 1 | | / | | Adverse events | |
| L leading to Leading to treatment. L | | | | | |
| 1.6a treatment 1.6a discontinuation, by | | leading to | | leading to treatment | |

| | T 10 10 10 10 | 1 | 1 1 |
|---|---|---|---|
| | discontinuation, by<br>system organ class,<br>preferred term and<br>maximum grade -<br>Phase I (Safety set) | | system organ class, preferred term and maximum grade - Phase I (Safety set) |
| Table 14.3.1-<br>1.6b | Adverse events leading to treatment discontinuation, by system organ class, preferred term and maximum grade - Phase II (Safety set) | Table 14.3.1-<br>1.6b | Adverse events leading to treatment discontinuation, by system organ class, preferred term and maximum grade - Phase II (Safety set) |
| Table 14.3.1-1.10a | Overview of<br>adverse events of<br>special interest -<br>Phase I (Safety set) | Table 14.3.1-1.10a | Overview of adverse<br>events of special<br>interest - Phase I<br>(Safety set) |
| Table 14.3.1-<br>1.10b | Overview of<br>adverse events of<br>special interest -<br>Phase II (Safety<br>set) | Table 14.3.1-<br>1.10b | Overview of adverse events of special interest - Phase II (Safety set) |
| Table 14.3.1-1.17a | All deaths, by<br>system organ class<br>and preferred term<br>- Phase I (Safety<br>set) | Table 14.3.1-<br>1.17a | All deaths, by system organ class and preferred term - Phase I (Safety set) |
| Table 14.3.1-<br>1.17b | All deaths, by<br>system organ class<br>and preferred term<br>- Phase II (Safety<br>set) | Table 14.3.1-<br>1.17b | All deaths, by system organ class and preferred term - Phase II (Safety set) |
| Table 14.3.1-1.19 | Non-serious<br>adverse events<br>(threshold = 5%)<br>by system organ<br>class and preferred<br>term for all<br>subjects (Safety<br>set) | Table 14.3.1-1.19 | Non-serious adverse<br>events (threshold =<br>5%) by system organ<br>class and preferred<br>term for all subjects<br>(Safety set) |
| Table 14.3.1-<br>1.21a | On-treatment<br>deaths and serious<br>adverse events with<br>fatal outcome -<br>Phase I (Safety set) | Table 14.3.1-<br>1.21a | On-treatment deaths<br>and serious adverse<br>events with fatal<br>outcome - Phase I<br>(Safety set) |
| Table 14.3.1-<br>1.21b | On-treatment<br>deaths and serious<br>adverse events with<br>fatal outcome -<br>Phase II (Safety<br>set) | Table 14.3.1-<br>1.21b | On-treatment deaths<br>and serious adverse<br>events with fatal<br>outcome - Phase II<br>(Safety set) |

| | | T | T = |
|---|---|---|---|
| | Tumor assessments | | Tumor assessments |
| Listing 14.2-1.1b | and responses per | Listing 14.2-1.1b | and responses per |
| | BIRC – Phase II | | BIRC – Phase II Full |
| | Full analysis set | | analysis set |
| | Progression-free | | Progression-free |
| Listing 14.2-1.2b | survival per BIRC | Listing 14.2-1.2b | survival per BIRC – |
| 21341119 1 112 1 12 1 | – Phase II Full | 2104119 1 1120 | Phase II Full analysis |
| | analysis set | | set |
| | Time to response | | Time to response and |
| | and duration of | | duration of response |
| Listing 14.2-1.3b | response per BIRC | Listing 14.2-1.3b | per BIRC – Phase II |
| | – Phase II Full | | Full analysis set |
| | analysis set | | , |
| | Tumor assessments | | Tumor assessments |
| - | and response per | | and response per |
| Listing 14.2-2.1a | investigator | Listing 14.2-2.1a | investigator |
| | assessment – Phase | | assessment – Phase I |
| | I Full analysis set | | Full analysis set |
| | Tumor assessments | | Tumor assessments |
| T: /: 140011 | and response per | T: 4: 140011 | and response per |
| Listing 14.2-2.1b | investigator | Listing 14.2-2.1b | investigator |
| | assessment – Phase | | assessment – Phase II |
| | II Full analysis set | | Full analysis set |
| | Progression-free | | Progression-free |
| T: /: 14000 | survival per | 1 14000 | survival per |
| Listing 14.2-2.2a | investigator | Listing 14.2-2.2a | investigator |
| | assessment – Phase | | assessment – Phase I |
| | I Full analysis set | | Full analysis set |
| | Progression-free | | Progression-free |
| Listing 14 2 2 2h | survival per investigator | Listing 14.2.2.2h | survival per investigator |
| Listing 14.2-2.2b | assessment – Phase | Listing 14.2-2.2b | assessment – Phase II |
| | II Full analysis set | | Full analysis set |
| | Time to response | | Tull allalysis set |
| | and duration of | | Time to response and |
| | response per | | duration of response |
| Listing 14.2-2.3a | investigator | Listing 14.2-2.3a | per investigator |
| | assessment – Phase | | assessment – Phase I |
| | I Full analysis set | | Full analysis set |
| | Time to response | | |
| | and duration of | | Time to response and |
| | response per | | duration of response |
| Listing 14.2-2.3b | investigator | Listing 14.2-2.3b | per investigator |
| | assessment – Phase | | assessment – Phase II |
| | II Full analysis set | | Full analysis set |
| T | Overall survival – | T1.1 11.0 0.1 | Overall survival – |
| Listing 14.2-2.6a | Phase I Safety set | Listing 14.2-2.6a | Phase I Safety set |
| T 1 1 1 1 1 2 2 2 2 | Overall survival – | T 11000 | Overall survival – |
| Listing 14.2-2.6b | Phase II Safety set | Listing 14.2-2.6b | Phase II Safety set |
| Listing 14.3.2- | Deaths - Phase I | Listing 14.3.2- | Deaths - Phase I |
| 1.1a | (Safety set) | 1.1a | (Safety set) |
| Listing 14.3.2- | Deaths - Phase II | Listing 14.3.2- | Deaths - Phase II |
| 1.1b | (Safety set) | 1.1b | (Safety set) |

| | 1 | 1 | |
|---|---|---|---|
| Listing 14.3.2- | Serious adverse | Listing 14.3.2- | Serious adverse |
| 2.1a | events - Phase I | 2.1a | events - Phase I |
| 2.1a | (Safety set) | 2.1a | (Safety set) |
| | Serious adverse | | Serious adverse |
| Listing 14.3.2- | events - Phase II | Listing 14.3.2- | events - Phase II |
| 2.1b | (Safety set) | 2.1b | (Safety set) |
| T 1 1 1 1 0 0 | Serious adverse | T | Serious adverse |
| Listing 14.3.2- | events with fatal | Listing 14.3.2- | events with fatal |
| 2.2a | outcome - Phase I | 2.2a | outcome - Phase I |
| | (Safety set) | | (Safety set) |
| | Serious adverse | | Serious adverse |
| Listing 14.3.2- | events with fatal | Listing 14.3.2- | events with fatal |
| 2.2b | outcome - Phase II | 2.2b | outcome - Phase II |
| | (Safety set) | | (Safety set) |
| | Adverse events | | Adverse events |
| Listing 14.3.2- | leading to | Listing 14.3.2- | leading to |
| 3.1a | discontinuation - | 3.1a | discontinuation - |
| 3.14 | | 3.1a | |
| | Phase I (Safety set) | | Phase I (Safety set) |
| | Adverse events | | Adverse events |
| Listing 14.3.2- | leading to | Listing 14.3.2- | leading to |
| 3.1b | discontinuation - | 3.1b | discontinuation - |
| 3.10 | Phase II (Safety | 3.10 | |
| | set) | | Phase II (Safety set) |
| | Adverse events | | Adverse events |
| | leading to dose | | leading to dose |
| Listing 14.3.2- | adjustment and/or | Listing 14.3.2- | adjustment and/or |
| 4.1a | | 4.1a | interruption - Phase I |
| | interruption - | | |
| | Phase I (Safety set) | | (Safety set) |
| | Adverse events | | Adverse events |
| | leading to dose | | leading to dose |
| Listing 14.3.2- | adjustment and/or | Listing 14.3.2- | adjustment and/or |
| 4.1b | interruption - | 4.1b | interruption - Phase |
| | Phase II (Safety | | |
| | set) | | II (Safety set) |
| | Adverse events of | | Adverse events of |
| Listing 14.3.2- | special interest - | Listing 14.3.2- | special interest - |
| 5.1a | Phase I (Safety set) | 5.1a | Phase I (Safety set) |
| | ` • | | Thase I (Salety set) |
| T '-4' 14 2 2 | Adverse events of | T '-4' 14 2 2 | Adverse events of |
| Listing 14.3.2- | special interest - | Listing 14.3.2- | special interest - |
| 5.1b | Phase II (Safety | 5.1b | Phase II (Safety set) |
| | set) | | ` ' ' |
| Listing 16.2.1- | Subject disposition | Listing 16.2.1- | Subject disposition - |
| _ | - Phase I (Full | _ | Phase I (Full analysis |
| 1.1a | analysis set) | 1.1a | set) |
| | Subject disposition | | Subject disposition - |
| Listing 16.2.1- | - Phase II (Full | Listing 16.2.1- | Phase II (Full |
| 1.1b | analysis set) | 1.1b | analysis set) |
| | Informed consent | | Informed consent |
| Listing 16.2.1- | | Listing 16.2.1- | |
| 1.3 | (All screened | 1.3 | (All screened |
| | subjects) | | subjects) |
| Listing 16.2.2- | Protocol deviations | Listing 16.2.2- | Protocol deviations - |
| 1.1a | - Phase I (Full | | Phase I (Full analysis |
| 1.1a | analysis set) | 1.1a | set) |
| | . , | 1 | / |

| | <b>T</b> | | |
|---|---|---|---|
| Listing 16.2.2-<br>1.1b | Protocol deviations - Phase II (Full | Listing 16.2.2-<br>1.1b | Protocol deviations - Phase II (Full |
| Listing 16.2.4-<br>1.3a | analysis set) Relevant medical history and current medical conditions - Phase I (Full analysis set) | Listing 16.2.4-<br>1.3a | analysis set) Relevant medical history and current medical conditions - Phase I (Full analysis set) |
| Listing 16.2.4-<br>1.3b | Relevant medical<br>history and current<br>medical conditions<br>- Phase II (Full<br>analysis set) | Listing 16.2.4-<br>1.3b | Relevant medical<br>history and current<br>medical conditions -<br>Phase II (Full<br>analysis set) |
| Listing 16.2.4-<br>1.7a | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Surgery - Phase I<br>(Full analysis set) | Listing 16.2.4-<br>1.7a | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug - Surgery<br>- Phase I (Full<br>analysis set) |
| Listing 16.2.4-<br>1.7b | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Surgery - Phase II<br>(Full analysis set) | Listing 16.2.4-<br>1.7b | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug - Surgery<br>- Phase II (Full<br>analysis set) |
| Listing 16.2.4-<br>1.8a | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Radiotherapy -<br>Phase I (Full<br>analysis set) | Listing 16.2.4-<br>1.8a | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Radiotherapy - Phase<br>I (Full analysis set) |
| Listing 16.2.4-<br>1.8b | Antineoplastic therapies since discontinuation of study drug - Radiotherapy - Phase II (Full analysis set) | Listing 16.2.4-<br>1.8b | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Radiotherapy - Phase<br>II (Full analysis set) |
| Listing 16.2.4-<br>1.9a | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Medications -<br>Phase I (Full<br>analysis set) | Listing 16.2.4-<br>1.9a | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Medications - Phase<br>I (Full analysis set) |
| Listing 16.2.4-<br>1.9b | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Medications -<br>Phase II (Full<br>analysis set) | Listing 16.2.4-<br>1.9b | Antineoplastic<br>therapies since<br>discontinuation of<br>study drug -<br>Medications - Phase<br>II (Full analysis set) |

| | 1 5 | 1 | |
|---|---|---|---|
| Listing 16.2.5-<br>1.1a | Dose<br>administration<br>record - Phase I<br>(Safety set) | Listing 16.2.5-<br>1.1a | Dose administration<br>record - Phase I<br>(Safety set) |
| Listing 16.2.5-<br>1.1b | Dose administration record - Phase II (Safety set) | Listing 16.2.5-<br>1.1b | Dose administration<br>record - Phase II<br>(Safety set) |
| Listing 16.2.7-<br>1.1a | Adverse events -<br>Phase I (Safety set) | Listing 16.2.7-<br>1.1a | Adverse events -<br>Phase I (Safety set) |
| Listing 16.2.7-<br>1.1b | Adverse events -<br>Phase II (Safety<br>set) | Listing 16.2.7-<br>1.1b | Adverse events -<br>Phase II (Safety set) |
| Listing 16.2.8-<br>1.1a | CTC grade 3 or 4<br>laboratory values -<br>Phase I (Safety set) | Listing 16.2.8-<br>1.1a | CTC grade 3 or 4<br>laboratory values -<br>Phase I (Safety set) |
| Listing 16.2.8-<br>1.1b | CTC grade 3 or 4<br>laboratory values -<br>Phase II (Safety<br>set) | Listing 16.2.8-<br>1.1b | CTC grade 3 or 4<br>laboratory values -<br>Phase II (Safety set) |
| Listing 16.2.8-<br>1.2a | Hematology -<br>primary<br>hematology<br>variables - Phase I<br>(Safety set) | Listing 16.2.8-<br>1.2a | Hematology -<br>primary hematology<br>variables - Phase I<br>(Safety set) |
| Listing 16.2.8-<br>1.2b | Hematology -<br>primary<br>hematology<br>variables - Phase<br>II (Safety set) | Listing 16.2.8-<br>1.2b | Hematology -<br>primary hematology<br>variables - Phase II<br>(Safety set) |
| Listing 16.2.8-<br>1.3a | Hematology -<br>WBC and<br>differentials -<br>Phase I (Safety set) | Listing 16.2.8-<br>1.3a | Hematology - WBC<br>and differentials -<br>Phase I (Safety set) |
| Listing 16.2.8-<br>1.3b | Hematology -<br>WBC and<br>differentials -<br>Phase II (Safety<br>set) | Listing 16.2.8-<br>1.3b | Hematology - WBC<br>and differentials -<br>Phase II (Safety set) |
| Listing 16.2.8-<br>1.4a | Hematology -<br>coagulation -<br>Phase I (Safety set) | Listing 16.2.8-<br>1.4a | Hematology -<br>coagulation - Phase I<br>(Safety set) |
| Listing 16.2.8-<br>1.4b | Hematology -<br>coagulation -<br>Phase II (Safety<br>set) | Listing 16.2.8-<br>1.4b | Hematology -<br>coagulation - Phase<br>II (Safety set) |
| Listing 16.2.8-<br>1.5a | Biochemistry -<br>liver - Phase I<br>(Safety set) | Listing 16.2.8-<br>1.5a | Biochemistry - liver<br>- Phase I (Safety set) |
| Listing 16.2.8-<br>1.5b | Biochemistry -<br>liver - Phase II<br>(Safety set) | Listing 16.2.8-<br>1.5b | Biochemistry - liver<br>- Phase II (Safety set) |

| Listing 16.2.8-<br>1.6a | Biochemistry -<br>renal - Phase I<br>(Safety set) | Listing 16.2.8-<br>1.6a | Biochemistry - renal -<br>Phase I (Safety set) |
|---|---|---|---|
| Listing 16.2.8-<br>1.6b | Biochemistry -<br>renal - Phase II<br>(Safety set) | Listing 16.2.8-<br>1.6b | Biochemistry - renal -<br>Phase II (Safety set) |
| Listing 16.2.8-<br>1.7a | Biochemistry -<br>other - Phase I<br>(Safety set) | Listing 16.2.8-<br>1.7a | Biochemistry - other<br>- Phase I (Safety set) |
| Listing 16.2.8-<br>1.7b | Biochemistry -<br>other - Phase II<br>(Safety set) | Listing 16.2.8-<br>1.7b | Biochemistry - other<br>- Phase II (Safety set) |
| Listing 16.2.8-<br>1.8a | Urinary<br>parameters:<br>urinalysis (dipstick<br>analysis) - Phase I<br>(Safety set) | Listing 16.2.8-<br>1.8a | Urinary parameters:<br>urinalysis (dipstick<br>analysis) - Phase I<br>(Safety set) |
| Listing 16.2.8-<br>1.8b | Urinary<br>parameters:<br>urinalysis (dipstick<br>analysis) - Phase II<br>(Safety set) | Listing 16.2.8-<br>1.8b | Urinary parameters:<br>urinalysis (dipstick<br>analysis) - Phase II<br>(Safety set) |
| Listing 16.2.8-<br>1.9a | Urinary parameters: urinalysis (microscopic analysis) - Phase I (Safety set) | Listing 16.2.8-<br>1.9a | Urinary parameters:<br>urinalysis<br>(microscopic<br>analysis) - Phase I<br>(Safety set) |
| Listing 16.2.8-<br>1.9b | Urinary<br>parameters:<br>urinalysis<br>(microscopic<br>analysis) - Phase II<br>(Safety set) | Listing 16.2.8-<br>1.9b | Urinary parameters:<br>urinalysis<br>(microscopic<br>analysis) - Phase II<br>(Safety set) |
| Listing 16.2.8-<br>1.10a | Subjects with worst post-baseline Total bilirubin > 2xULN and AT > 3xULN values - Phase I (Safety set) | Listing 16.2.8-<br>1.10a | Subjects with worst post-baseline Total bilirubin > 2xULN and AT > 3xULN values - Phase I (Safety set) |
| Listing 16.2.8-<br>1.10b | Subjects with worst post-baseline Total bilirubin > 2xULN and AT > 3xULN values - Phase II (Safety set) | Listing 16.2.8-<br>1.10b | Subjects with worst post-baseline Total bilirubin > 2xULN and AT > 3xULN values - Phase II (Safety set) |
| Listing 16.2.8-<br>1.11a | Subject laboratory<br>profile of hepatic<br>laboratory values -<br>Phase I (Safety set) | Listing 16.2.8-<br>1.11a | Subject laboratory<br>profile of hepatic<br>laboratory values -<br>Phase I (Safety set) |
| Listing 16.2.8-<br>1.11b | Subject laboratory profile of hepatic laboratory values - | Listing 16.2.8-<br>1.11b | Subject laboratory profile of hepatic |

| | Phase II (Safety set) | | laboratory values -<br>Phase II (Safety set) | |
|---|---|---|---|---|
| Listing 16.2.9-<br>1.1a | Notable vital sign<br>values - Phase I<br>Safety set | Listing 16.2.9-<br>1.1a | Notable vital sign<br>values - Phase I<br>Safety set | |
| Listing 16.2.9-<br>1.1b | Notable vital sign<br>values - Phase II<br>Safety set | Listing 16.2.9-<br>1.1b | Notable vital sign<br>values - Phase II<br>Safety set | |
| Listing 16.2.9-<br>1.2a | Vital signs - Phase<br>I Safety set | Listing 16.2.9-<br>1.2a | Vital signs - Phase I<br>Safety set | |
| Listing 16.2.9-<br>1.2b | Vital signs - Phase<br>II Safety set | Listing 16.2.9-<br>1.2b | Vital signs - Phase II<br>Safety set | |
| Listing 16.2.9-<br>2.1a | Notable ECG<br>values - Phase I<br>Safety set | Listing 16.2.9-<br>2.1a | Notable ECG values - Phase I Safety set | |
| Listing 16.2.9-<br>2.1b | Notable ECG<br>values - Phase II<br>Safety set | Listing 16.2.9-<br>2.1b | Notable ECG values - Phase II Safety set | |
| Listing 16.2.9-<br>2.2a | ECG values -<br>Phase I Safety set | Listing 16.2.9-<br>2.2a | ECG values - Phase I<br>Safety set | |
| Listing 16.2.9-<br>2.2b | ECG values -<br>Phase II Safety set | Listing 16.2.9-<br>2.2b | ECG values - Phase<br>II Safety set | |
| Listing 16.2.9-<br>3.1a | Pregnancy test<br>results - Phase I<br>Safety set | Listing 16.2.9-<br>3.1a | Pregnancy test results - Phase I Safety set | |
| Listing 16.2.9-<br>3.1b | Pregnancy test<br>results - Phase II<br>Safety set | Listing 16.2.9-<br>3.1b | Pregnancy test results - Phase II Safety set | |
| Listing 16.2.9-5.1a | Hepatitis screen<br>and monitoring -<br>Phase I Safety set | Listing 16.2.9-<br>5.1a | Hepatitis screen and<br>monitoring - Phase I<br>Safety set | Please change column title "Hepatitis screen" to "Hepatitis assessment" |
| Listing 16.2.9-<br>5.1b | Hepatitis screen<br>and monitoring -<br>Phase II Safety set | Listing 16.2.9-<br>5.1b | Hepatitis screen and<br>monitoring - Phase II<br>Safety set | |